CLINICAL TRIAL: NCT00541606
Title: Pharmacist Assisted Medication Program Enhancing the Regulation of Diabetes (PAMPERED)
Brief Title: Pharmacist Assisted Medication Program Enhancing the Regulation of Diabetes
Acronym: PAMPERED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahey Clinic (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PAMPERED
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Pharmaceutical Care; Collaborative Practice
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Received collaborative care including a clinical pharmacist practitioner.
  Interventions: Other: Pharmacist collaboration in diabetes care
- Control (Active Comparator): Patients received usual care directed by their physician.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Pharmacist collaboration in diabetes care — Patients attended a minimum of 3 clinic visits (month 0, 6, 12) with one of the clinical pharmacists, where targeted physical assessment, education, and medication changes and follow up were recommended. Additional visits were arranged as clinically appropriate for drug monitoring. Referrals were facilitated to other clinicians where indicated, including ophthalmology, podiatry, CDEs, nutrition, and primary care. The pharmacists' recommendations for medication adjustment, laboratory monitoring and referrals were based upon the most recent guidelines and clinical trial evidence. Any therapy adjustment, lab testing or referrals required approval by the referring physician. A1c, lipid and BP values were collected prospectively at months 0, 6 and 12.
  Arms: Intervention
Other: Usual care — Control patients received usual care directed by their physician, and the same data were gathered from chart review during the 12-month study period.
  Arms: Control

SUMMARY:
The purpose of this study is to demonstrate that pharmacists working collaboratively with physicians and other providers in an ambulatory care setting can improve glucose, blood pressure, and lipid control, as well as improve quality of life, adherence to screening and general preventative measures.

DETAILED DESCRIPTION:
It is evident that a multi-disciplinary approach is key to the success in controlling the disease of diabetes and its complications. The value of pharmacists' involvement in disease state management in producing positive outcomes for patients has been well documented in the literature. There have been several studies that have shown that pharmacists' involvement in diabetes care improves glycemic control. There are also studies that look at pharmacists' management of glycemic control and adherence to the ADA guidelines. Many of these studies are retrospective, lack a randomized control group, had a small study sample, or were short term. We undertook a prospective, randomized study to demonstrate that pharmacists working collaboratively with physicians and other providers in an ambulatory care setting can improve glucose, blood pressure, and lipid control, as well as improve quality of life, adherence to screening and general preventative measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* A1c > 8% within the 6 months prior to the data acquisition date
* Primary Care physician at Lahey Clinic Burlington site
* Diagnosis of T2 DM for minimum of 6 months

Exclusion Criteria:

* Concurrently enrolled in any other pharmacist-run or diabetes study
* Receiving diabetes management by an outside provider
* A medical condition that may adversely affect compliance with the treatment protocol

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2000-09; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Primary outcomes included the achievement of targets for A1c (< or = 7%), LDL cholesterol (< or = 100 mg/dL) and blood pressure (< or = 130/80), changes in quality of life as measured by the SF-36 Health Survey, and patient satisfaction. | 12 months

SECONDARY OUTCOMES:
Secondary outcomes included diabetes-related hospitalizations and acute care visits during the study period for both the intervention and control groups. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary Cushing, MD, Principal Investigator — Lahey Clinic, Burlington, MA; Michelle Jacobs, PharmD, Study Director — Currently: Northeastern University, Boston, MA
Locations (1):
- Lahey Clinic, Burlington, Massachusetts, United States